CLINICAL TRIAL: NCT03203785
Title: Effect of Carbohydrate Consumption on Fatigue and Muscle Damage in Jiu-Jitsu Athletes: A Randomized Clinical Trial
Brief Title: Effect of Carbohydrate Consumption on Fatigue and Muscle Damage in Jiu-Jitsu Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Cláudia Dornelles Schneider, Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 1.873.861
Record Dates: First submitted 2017-06-26; First posted 2017-06-29 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Fatigue; Exercise-induced Muscle Damage
MeSH Terms: conditions — Fatigue | interventions — Carbohydrates; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate (Experimental): 30g of carbohydrate (maltodextrin) diluted in 300ml of water. Athletes will drink 100ml before and 100ml in the first and second interval between exercise.
  Interventions: Dietary Supplement: Carbohydrate (maltodextrin)
- Placebo (Placebo Comparator): 300 ml of a non-caloric drink. Athletes will drink 100ml before and 100ml in the first and second interval between exercise.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Carbohydrate (maltodextrin) — maltodextrin flavored
  Arms: Carbohydrate
Other: Placebo — non-caloric drink
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blinded, placebo-controlled trial that will include the participation of 14 Jiu-Jitsu athletes between 18 and 33 years. The aim of the study is to evaluate the effects of carbohydrate consumption on fatigue and exercise-induced muscle damage in Jiu-Jitsu athletes.

DETAILED DESCRIPTION:
Brazilian Jiu-Jitsu (BJJ) is a sport characterized by intermittent high-intensity efforts separated by periods of low intensity. Muscular strength is considered one of the most important physical components to be developed, especially in the upper limbs through dynamic and static actions. The activities of high intensity (relation effort-pause) carried out by the upper and lower limbs during BJJ can induce muscle fatigue. In order to minimize the glycogen depletion and to guarantee the availability of energy substrate to the athlete during the physical exercise, the carbohydrate intake before moderate intensity exercises should be between 5-7 g / kg of weight / day. The intervention group will receive a 30g maltodextrin beverage and the placebo group a non-carbohydrate drink. There will be 3 combat simulations of 8 min each, with intervals of 10 min between fights. Athletes will be instructed to remain with their usual intake during the study. The outcomes will be: manual grip strength (dynamometer), upper limb strength (KGST), lower limb strength (vertical jump), subjective exertion perception (Borg scale), pain perception (Nilsson scale), blood markers of muscle damage (CK and LDH), lactate, and glycemia.

ELIGIBILITY:
Inclusion Criteria:

* Compete in the categories of weight between 70kg and 88,3kg (weight classification from light to medium heavy, belonging to the bands purple to brown).
* Age between 18 and 33 years.
* Be training at least three times a week, minimum of 1,5 hours per day, for at least 3 consecutive months.
* Have not used anabolic steroids in the last 6 months during the study period.
* Do not use any type of dietary supplement in the last 3 months.
* Self-declared healthy individuals.

Exclusion Criteria:

* Recent muscle injury (within the last 3 months) that compromises and / or impedes the performance of the exercise requested in the study.
* Be in a time of rapid weight loss (pre-competition).

Ages: 18 Years to 33 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
change in upper limbs strength | Pre-exercise; at 2 intervals during exercise; 24hour and 48hour after exercise
  Kimono Grip Strength Test

SECONDARY OUTCOMES:
change in lower limbs power | Pre-exercise; at 2 intervals during exercise; 24hour and 48hour after exercise
  Horizontal Countermovement Jump
change in hand grip strength | Pre-exercise; at 2 intervals during exercise; 24hour and 48hour after exercise
  Grip Strength Test
change in creatine kinase | Pre-exercise; immediatly post-exercise; 24hour and 48hour after exercise
  3 ml of blood samples
change in glucose | Pre-exercise; at 2 intervals during exercise; immediatly post-exercise
  fingertip blood measured by Accutrend® Active glucose-specific reagent tape
change in lactate | At 2 intervals during exercise; immediatly post-exercise
  fingertip blood measured by Accutrend Plus.
change in lactate dehydrogenase | Pre-exercise; immediatly post-exercise; 24hour and 48hour after exercise
  3 ml of blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Claudia D Schneider, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Gabriella B. Möller, Pôrto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided